CLINICAL TRIAL: NCT00305071
Title: A Double-Blind, Randomized, Placebo-Controlled Study to Evaluate the Effect of Adjuvant Treatment With Compound Cranberry Extract Tablets (UmayC) in Acute Bacterial Cystitis.
Brief Title: Effect of Adjuvant Treatment With Compound Cranberry Extract Tablets in Acute Bacterial Cystitis.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Min-Sheng General Hospital (Other)
Collaborators: Acrobio Healthcare Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ICMJE IRB NO：950113-1
Record Dates: First submitted 2006-03-19; First posted 2006-03-21 (Estimated); Last update posted 2006-03-21 (Estimated); Status verified 2006-03

CONDITIONS: Pyuria; Urinary Tract Infections
Keywords: pyuria; urinary tract infections; Vaccinium macrocarpon
MeSH Terms: conditions — Pyuria; Urinary Tract Infections

INTERVENTIONS:
Drug: compound cranberry extract tablet

SUMMARY:
In conventional treatment for non-complicated bacterial cystitis, 3-day oral antibiotics could achieve good cure rate. However, severe lower urinary tract symptoms were most bothersome and only could be partially relieved by NSAID, detrusor muscle relaxants, minor tranquilizer or pyridium. Some medication associated side effects were complained while receiving adjuvant medication treatment, including gastro-intestinal discomfort, dry mouth, blurred vision, lethargy, or allergic reactions. The irritative bladder symptoms from bladder inflammation had great impact on the quality of life and well tolerable adjuvant therapy would have clinical benefit to reduce the discomfort from the bladder.

In the past years, cranberry juice or its extract has been proven to have protective effect on urothelium to prevent further bacterial ascending infection. The commercial cranberry extract tablets have good tolerability and showed good effect on symptoms reliving and infection protection on several clinical observation. In acute bladder infection, we could expect the bioactive components in cranberry could reduce the virulence of pathogens and assist to eradicate pathogens and to stable the urothelium. In literature review, only little works focusing on the symptoms relief in acute cystitis patients. To clarify the clinical benefit on lower urinary symptoms relieving, we attempt to conduct a randomized double-blind placebo-controlled trial to evaluate the effect of a compound cranberry extract tablet as an adjunctive modality in treating acute uncomplicated bacterial cystitis in otherwise healthy female patients.

DETAILED DESCRIPTION:
Introduction

Acute bacterial cystitis is a common and bothersome disease with a rapid onset nature. Uncomplicated cystitis occurs in patients without anatomical or physiological anomaly in the lower urinary tract. Although the infection is not life threatening in immuno-competent patients, the associated lower urinary tract symptoms cause massive impact on the quality-of-life of the victims. The voiding symptoms, such as urinary frequency, urgency, dysuria and suprapubic pain, were associated with the inflammatory response to microbial invasion. In most clinical scenario, 3-day empirical oral antimicrobial treatment could eradicate the pathogen efficiently.1,2 However, the lower urinary tract symptoms were not eradicated effectively by antibiotics only. In daily clinical practice, several symptomatic relieving treatments were applied while acute infection presented, including pyridine and anticholinergic agents. However, several side effects were complained according to the medication.

In lower urinary tract infection, the virulence of the pathogen was the major factor associated with colonization and invasion in the urinary tract mucosa. The adherence of the pathogen to the urothelium is the crucial step in the urinary tract infection.3 Several studies revealed good anti-adherence effect of the cranberry juice.4-7 In several clinical studies, cranberry juice has been proven to be an protective effect in bacterial cystitis8 and the role of cranberry juice in preventing urinary tract infection was well established.9,10 Cranberry is a rich source of bioactive compounds, such as phenolic acid and several organic acids, which have been proven playing major anti-bacterial effect.11

In literature reviewing, the clinical application of cranberry juice or extract tablet was focusing on the preventive role on chronic or repeated urinary tract infection. The effect to reduce bacteriuria and pyuria has been mentioned.12 However, the effect on lower urinary tract symptom relieving effect of the food supplement cranberry was not established. In this study, we try to evaluate the clinical efficacy of a commercial compound cranberry extract in treating acute uncomplicated cystitis as an adjunctive role. The compound tablet contained 900mg per tablet, including 600% concentrated cranberry extract 150mg, vitamin C 70mg, Rhizoma extract (Acrobio TS®) 150mg, Flos extract (Acrobio GL®) 60mg, lactose and mannitol 490mg. The compound has been on the market in Taiwan as a food supplement and was well tolerable. We conducted a double-blind, randomized, placebo-controlled trial to evaluate the adjuvant effect of compound cranberry extract on the symptomatic relieving effect.

Material and Methods

Study Method:

We prepare to conduct a paralleled-group, double-blind, placebo-controlled, randomized clinical trial to evaluate the effect of a compound cranberry extract tablet as an adjunctive modality in treating acute uncomplicated bacterial cystitis in otherwise healthy female patients. The treatment arm will receive standard 3-day oral antibiotics plus 7-day compound cranberry extract tablets (UmayC) and the control arm will receive standard 3-day oral antibiotics plus 7-day identical placebo.

Study Processes:

1. Participant recruitment During study period, we will recruit 60 volunteer female patients visiting the urological outpatient clinics in Min-Sheng General Hospital for uncomplicated acute bacterial cystitis to join our trial. The age limitation was 20 to 65 years old and the acute cystitis was diagnosed by the clinical symptoms, physical exams and pyuria (WBC>5/HPF) on urinalysis.

   The exclusion criteria: recent (less than one month) urinary tract infection or partially treated acute cystitis; anatomical or function disease of the lower urinary tract; patients received radical pelvic surgery; associated bladder stone disease; upper urinary tract anomaly or urolithiasis; systemic infection with body temperature higher than 38°C; known allergic reaction to cranberry or vitamin C; pregnant or prepare to be pregnant, or diabetic patients.
2. Objectives and outcome measurements We try to evaluate the symptom relieving effect of compound cranberry extract as an adjuvant therapeutic modality. The study hypothesis is the compound cranberry extract tablet as an adjuvant treatment for uncomplicated acute bacterial cystitis with 3-day empirical antibiotics will reduce the irritative bladder symptoms (urinary frequency, urinary urgency, and dysuria and suprapubic pain).

   We conducted a Frequency-Urgency-Pain (FUP) score to evaluate the irritative lower urinary tract symptoms. Another 10-point Likert scales from 0 (none) to 9 (severe) questionnaire will be used to evaluate every individual symptom. A modified diary method was used to evaluate the symptoms change during the whole evaluation period. 3 in-face questionnaire interviews will be preformed on day 1, 4, and 8 by the study assistants. A brief form questionnaire will be done by telephone on day 2 and 3. The primary outcome of this study is the proportion of symptoms relief (based on FUP and individual symptom scale evaluation) after 3-day and 7-day treatments. The secondary outcome variables were the pyuria eradication rate after 3- and 7-day therapy and the time to symptoms relief. Possible adverse effect was recorded and reported.
3. Sample size and randomization In this study, we will recruit 60 participants to detect the difference between the intervention and control groups with a 0.05 one-sided significance level and a 80% power. These participants will be randomly assigned to each group according to a pre-set random permuted blocks procedure. Efficacy analysis will be conducted according to the intension-to-treat principle.
4. Intervention Intervention group will receive 3-day oral trimethoprim/sulfamethoxazole (80/400mg) 2 tablets twice a day on day 1 to 3 plus oral compound cranberry extract tablets (UmayC, 900mg) 2 tablets three times a day on day 1 to 7. The control group will received same oral antibiotics plus identical placebo prescribed as the same protocol of intervention arm. For patients with known allergic reaction to sulfa drug, the empirical antibiotics will be replaced by cephalexin (250mg) 2 capsules four times a day.

Study Processes:

After participant enrollment with inform consent, detail medical history will be collected, including basic physiological data (body weight and height), major medical disease (diabetes, cerebral vascular disease, or neurological disorder), major operation history (neurological and pelvic surgery), recent medication records (including recent antibiotics treatment), child-baring history, sexual activity, fluid drinking history, and socio-economical and education status.

A voiding symptoms questionnaire, including FUP score and 10-point Likert scales symptomatic questions, will be done by in-face interview by study assistants. Random urine bacterial culture will be collected before medical treatment. The participants will be requested to receive 2 telephone interviews on day 2 and 3 by the study assistants and to return for urinalysis and 2nd in-face questionnaire on day 4 after complete antibiotics treatment. The clinical follow up will be arranged on day 8 by the physicians and urinalysis will be done again.

Adverse event reporting and patient safety All participants will receive close follow up protocol for adverse event reporting. Any discomfort associated with the medical treatment will be recorded on daily interview record and be reported. Interruption of the trial and intervention decoding will be performed immediately once an intolerable side effect happened.

ELIGIBILITY:
Inclusion Criteria:

* female patient with non-complicated acute bacterial cystitis

Exclusion Criteria:

* recent (less than one month) urinary tract infection
* partially treated acute cystitis
* anatomical or function disease of the lower urinary tract
* patients received radical pelvic surgery
* associated bladder stone disease
* upper urinary tract anomaly or urolithiasis
* systemic infection with body temperature higher than 38°C
* known allergic reaction to cranberry or vitamin C
* pregnant or prepare to be pregnant.

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2006-04

PRIMARY OUTCOMES:
Time to symptoms relief

SECONDARY OUTCOMES:
Pyuria eradication rate

CONTACTS AND LOCATIONS:
Overall Officials: Po-Chien Huang, MD, Principal Investigator — Division of Urology, department of Surgery, Min-Sheng General Hospital, Taoyuan, Taiwan
Locations (1):
- Min-Sheng General Hospital, Taoyuan, Taiwan

REFERENCES:
- [Derived] Jepson RG, Mihaljevic L, Craig JC. Cranberries for treating urinary tract infections. Cochrane Database Syst Rev. 2023 Dec 14;12(12):CD001322. doi: 10.1002/14651858.CD001322.pub2. PMID 38096261